CLINICAL TRIAL: NCT07026474
Title: Randomized Phase III Trial of Sequential Re-Radiochemotherapy and Pembrolizumab Versus Immuno(Chemo)Therapy for Locoregionally Recurrent PD-L1 Positive HNSCC (CPS≥1)
Brief Title: Re-Radiochemotherapy and Pembrolizumab vs. Immuno(Chemo)Therapy for Locoregionally Recurrent PD-L1 Positive (CPS≥1) HNSCC
Acronym: RePaIr-HN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RePaIr-HN; 2024-520264-33-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy; Cisplatin; pembrolizumab; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational arm (Experimental): Patients receive Re-RCT followed by pembrolizumab immunotherapy for up to 2 years. Concomitant chemotheraphy is cisplatin. In case of renal dysfunction cisplatin can be switched to carboplatin.
  Interventions: Other: radiotherapy; Drug: Cisplatin; Drug: Alternative medications: carboplatin; Drug: Pembrolizumab
- Control arm (Active Comparator): Patients receive pembrolizumab monotherapy for up to 2 years. At the discretion of the treating physician, up to 6 additional cycles of cisplatin or carboplatin in combination with 5-fluorouracil may be given.
  Interventions: Drug: Pembrolizumab; Drug: cisplatin + 5-fluorouracil (5FU); Drug: Alternative medications: carboplatin + 5-fluorouracil (5FU)

INTERVENTIONS:
Other: radiotherapy — single doses of 1.8Gy up to a total dose of 55.8Gy to 63.0Gy
  Arms: Investigational arm
Drug: Cisplatin — 40mg/m² BSA weekly concomitant to re-irradiation
  Arms: Investigational arm
Drug: Pembrolizumab — i.v., 200mg absolute, q3w
  Arms: Control arm
Drug: cisplatin + 5-fluorouracil (5FU) — Cisplatin: 100mg/m² BSA d1, q3w / 5-FU: 1000mg/m² BSA d1-4, q3w
  Arms: Control arm
Drug: Alternative medications: carboplatin + 5-fluorouracil (5FU) — Carboplatin: AUC5 d1, q3w / 5-FU: 1000mg/m² BSA d1-4, q3w
  Arms: Control arm
Drug: Alternative medications: carboplatin — AUC2 weekly
  Arms: Investigational arm
Drug: Pembrolizumab — i.v., 200mg absolute, q3w, starting within 8-14 days after completion of RCT
  Arms: Investigational arm

SUMMARY:
Prospective, open-label, randomized controlled phase III trail that aims to investigate whether Re-Radiochemotherapy (Re-RCT) and sequential immunotherapy with pembrolizumab improves overall survival compared to the standard treatment with pembrolizumab alone (± chemotherapy) in locoregionally recurrent PD-L1 positive (CPS≥1) HNSCC.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the subject prior to performing any protocol-related procedures.
* Age ≥ 18 years at time of study entry.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Locoregionally recurrent or second primary HNSCC.
* Histological confirmation of HNSCC.
* Tumor is surgically not resectable or surgical resection bears great potential for relevant functional morbidity or patient refuses surgery.
* No distant metastases (cM0).
* PD-L1 combined positive score (CPS) ≥1 according to local pathological PD-L1 assessment. A validated test must be used in an accredited laboratory.
* Prior radio(chemo)therapy of the neck (time interval ≥ 6 months).
* Adequate normal organ and marrow function as defined: Haemoglobin ≥ 9.0 g/dL; Leukocytes (WBC) ≥ 3,000 per mm3or Neutrophils ≥ 1,500 per mm3; Platelet count > 100,000 per mm3.
* Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of haemolysis or hepatic pathology).
* AST (SGOT) / ALT (SGPT) ≤ 2.5 x institutional ULN.
* Creatinine Clearance ≥ 40ml/min (calculated from serum creatinine using the Cockcroft-Gault formula).
* Female subject of childbearing potential should have a negative serum pregnancy within 72 hours prior to receiving the first dose of RT and/or the first dose of pembrolizumab. A highly sensitive pregnancy test must be used.
* Female subjects of childbearing potential must be willing to use a highly effective contraceptive measure (see also Section 7.1.9 Contraception and pregnancy testing during the trial). Highly effective contraception is required for the course of the trial through 120 days after the last dose of trial therapy.
* Generative male subjects must agree to use a highly effective method of contraception (see also Section 7.1.9 Contraception and pregnancy testing during the trial), starting with the first dose of trial therapy through 120 days after the last dose of trial therapy.
* Subject is willing and able to comply with the protocol for the duration of the trial including undergoing treatment and scheduled visits and examinations including.

Exclusion Criteria:

* Prior radio(chemo)therapy of the neck less than 6 months ago.
* Distant metastases (cM1).
* Is currently participating and receiving trial therapy or has participated in a trial of an investigational agent and received trial therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of trial treatment. The following are exceptions to this criterion:

  1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* Prior chemotherapy or targeted small molecule therapy within 2 weeks or anti-cancer monoclonal antibody (mAb) within 4 weeks prior to trial day 1 or who has not recovered from AEs due to a previously administered agent. (Subjects with ≤ grade 2 neuropathy are an exception to this criterion and may qualify for the trial.)
* History or concurrent other malignancy. Exceptions include patients, who have been disease free for at least 3 years. Further exceptions are completely resected basal cell carcinoma or squamous cell carcinoma of the skin or successfully treated in situ carcinoma.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* History of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has an active or chronic infection requiring systemic antibacterial, antifungal or antiviral therapy within 14 days prior to randomization or first dose of study drugs.
* Known hypersensitivity to the active substances or to any of the excipients.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Infection with human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
* Active hepatitis B (e.g., HBsAg reactive) or hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Live vaccine within 30 days of planned start of trial therapy.
* Performance status of >2 on the ECOG Performance Scale.
* Prior treatment with a PD-1/PD-L1 antibody in primary treatment of locally advanced HNSCC less than 6 months ago.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 2 years
  To evaluate the efficacy of a sequential treatment of Re-RCT followed by pembrolizumab compared to standard therapy with pembrolizumab ± chemotherapy, the primary endpoint of the trial is overall survival rate at 2 years.

CONTACTS AND LOCATIONS:
Locations (18):
- Germany (18):
  - Klinikum Chemnitz gGmbH, Klinik für Radioonkologie, Chemnitz
  - Klinikum Darmstadt GmbH, Institut für Radioonkologie und Strahlentherapie, Darmstadt
  - Gemeinschaftspraxis Hämatologie-Onkologie Dresden, Dresden
  - Uniklinikum Erlangen, Strahlenklinik, Erlangen
  - Universitätsmedizin Frankfurt, Klinik für Strahlentherapie und Onkologie, Frankfurt am Main
  - UKGM Gießen, Klinik für Strahlentherapie, Giessen
  - Universitätsklinikum Hamburg-Eppendorf, Zentrum für Onkologie; II. Medizinische Klinik und Poliklinik, Hamburg
  - Medizinische Hochschule Hannover (MHH), Klinik für Hämatologie, Hämostaseologie, Onkologie und Stammzelltransplantation, Hanover
  - Marien Hospital Herne, Klinik für Strahlentherapie und Radio-Onkologie, Herne
  - Universitätsklinikum des Saarlandes, Klinik für Strahlentherapie und Radioonkologie, Homburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Klinik und Poliklinik für Radioonkologie der Strahlentherapie, Mainz
  - Universitätsklinikum Münster, Klinik für Strahlentherapie - Radioonkologie, Münster
  - Universitätsklinikum Regensburg, Klinik und Poliklinik für Strahlentherapie, Regensburg
  - CaritasKlinikum Saarbrücken St. Theresia, Klinik für Radioonkologie und Strahlentherapie, Saarbrücken
  - Klinikum St.-Elisabeth Straubing GmbH, Klinik für Hals-Nasen-Ohren-Heilkunde, Straubing
  - Klinikum Stuttgart, Klinik für Strahlentherapie und Radioonkologie, Stuttgart
  - Universitätsklinikum Tübingen, Klinik für Radioonkologie, Tübingen
  - Universitätsklinikum Ulm, Klinik für Hals- Nasen-Ohrenheilkunde, Kopf- und Halschirurgie, Ulm

IPD SHARING:
Plan to Share IPD: No